CLINICAL TRIAL: NCT06003166
Title: Pharmaco-Diagnostic Crossover Trial for Peripheral Nerve Continuity After Trauma
Brief Title: 4-AP Peripheral Nerve Crossover Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, John Elfar, Tenured Professor, Chairman, Department of Orthopaedic Surgery, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 00002665; R01NS111293 (NIH)
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Nerve Injury; Crush Injury
Keywords: 4 aminopyridine; peripheral nerve; crush injury
MeSH Terms: conditions — Peripheral Nerve Injuries; Crush Injuries | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 4AP then placebo (Group A) (Experimental): Subjects randomized to this group will receive the study drug (4AP) followed by the placebo.
  Interventions: Drug: 4-Aminopyridine; Other: Placebo
- Placebo then 4AP (Group B) (Experimental): Subjects randomized to this group will receive the placebo first followed by the study drug (4AP)
  Interventions: Drug: 4-Aminopyridine; Other: Placebo

INTERVENTIONS:
Drug: 4-Aminopyridine — Study drug will be a one time, 10mg dose of 4-aminopyridine
  Other Names: 4AP
Other: Placebo — Matched placebo

SUMMARY:
The purpose of this study is to evaluate the role of single dose 4-aminopyridine (4-AP) on the diagnosis of severing vs non-severing nerve injury after peripheral nerve traction and/or crush injury. The investigational treatment will be used to test the hypothesis that 4-aminopyridine can speed the determination of nerve continuity after peripheral nerve traction and/or crush injuries allowing the identification of incomplete injuries earlier than standard electrodiagnostic (EDX) and clinical assessment.

Participants will be randomized to one of two groups to determine the order of treatment they receive (drug and placebo vs placebo and drug). Participants will undergo baseline testing for nerve assessment, receive either drug or placebo based on randomization and undergo hourly sensory and motor evaluation, EDX testing and serum 4AP levels for three hours after dosing. Participants will then repeat this with the crossover arm.

DETAILED DESCRIPTION:
This is a single-center study that will be conducted at the University of Arizona College of Medicine, Tucson. It is a double-blind, randomized, crossover trial design. Group A will receive the study drug followed by the placebo on the main trial day, and Group B will receive placebo first followed by the study drug. These groups will exist for both aims (both types of included patients).

Patients are randomized for the order (drug and placebo vs placebo and drug) of treatment they receive. Eligible, consented patients will present for testing from one of three locations (emergency department, inpatient ward, or home). Patients will undergo testing under the direction of trial personnel. Patients will undergo a thorough baseline sensory and motor evaluation and establish an intravenous line for blood sampling. A baseline blood sample (prior to drug and placebo) will be performed. These tests comprise part of a standardized array of tests performed hourly. This array of tests (serum 4AP level and sensorimotor examination) will be repeated every hour after treatment for three hours during which the drug will have decreased to a level low enough to have no expected effect. The final hourly test is the return to baseline test. It is likely going to occur at the third hourly post-test, but is depicted separately for clarity. Only three tests after dosing will be necessary, based on our expectations from known pharmacokinetic data. Patients will then repeat this with the crossover arm (drug vs placebo). Testing is concluded at the end of this period.

Following the initial testing, subjects will be seen for a period of 20 weeks after injury to monitor recovery and progress. Subjects will return for follow-up visits at 2, 6, 12, 18, and 20 weeks post injury. Subjects will receive a physical exam at all follow-up visit. Subjects will complete a telephone interview at 9 and 15 weeks post injury at which time subjective motor and sensory function will be assessed by asking 1) Can you move your (affected extremity)? Yes or No 2) Can you feel your (affected extremity)? Yes or No. Review of the subject diary will also be completed. The 9, 15, and 20 week visits are not part of standard of care and are being done for research purposes only. Each visit or phone interview will last approximately 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with trauma involving two or less limbs where the continuity of a given peripheral nerve or nerves is unclear on presenting physical examination.
* Closed soft tissue envelope obscuring direct observation of the continuity of the affected nerve.
* Cognitive ability to report sensory and motor deficit during examination.
* Eligible for standard of care plan of monitoring vs surgical exploration of the nerve.
* Adults subject aged 18-90
* Known limb trauma which resulted in nerve injury (aim 1) or post-operative/post intervention nerve injury (aim 2).
* Ability to give written informed consent.
* Availability for all testing days and main trial day.

Exclusion Criteria:

* Distracting injury which prevents adequate examination.
* Plan for surgical exploration of the nerve during the ensuing 48 hours.
* Plan for surgical exploration of the nerve as part of another surgical procedure within 48 hours of evaluation.
* Intoxication during examination or evidence of cognitive deficit that emerges during examination.
* History of multiple sclerosis, stroke or any other diagnosed neurological disorder
* History of hypersensitivity to AMPYRA® or 4-aminopyridine
* Current use of aminopyridine medications, including other compounded 4-AP
* Renal impairment based on calculated GFR (GFR<80 mL/min). This laboratory value is measured in all inpatient trauma patients as part of the standard of care.
* History of difficult compliance with timely follow up or plan to seek care at another institution closer to home.
* Patients outside the age range or unable to consent.
* Patients with a known history of a seizure disorder (4AP overdose can, in selected cases, result in limited seizure activity).
* Patients with a concomitant traumatic brain injury.
* Patients unable to communicate return or loss of sensation.
* Patients unable to exhibit motor control on the affected limb at baseline.
* Patients unwilling to complete the study requirements.
* Patients with injuries too extensive to isolate a single nerve(s) for testing.
* Patients currently taking organic cat-ion transporter 2 (OCT2) inhibitors, e.g. Cimetidine.
* Pregnancy, breastfeeding or incarcerated individuals.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Subjective return of sensation | During dosing of drug intervention and 2, 6, 9, 12, 15, 20 weeks post injury
  Return of lost sensation after nerve injury attributable to circulating 4AP. Subjective return of sensation in the injured limb or portion of the limb.
  Patients for this trial are not able to sense in portions of their limbs. The measure will be sensation, measured on the binary scale of yes or no (able to feel the extremity versus unable to feel). This is assessed through clinical examination of the injured limb.

CONTACTS AND LOCATIONS:
Overall Officials: John Elfar, MD, Principal Investigator — University of Arizona
Locations (1):
- Banner University Medical Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robinson LR. Role of neurophysiologic evaluation in diagnosis. J Am Acad Orthop Surg. 2000 May-Jun;8(3):190-9. doi: 10.5435/00124635-200005000-00006. PMID 10874226
- [Background] Robinson LR. Traumatic injury to peripheral nerves. Muscle Nerve. 2000 Jun;23(6):863-73. doi: 10.1002/(sici)1097-4598(200006)23:63.0.co;2-0. PMID 10842261
- [Background] Lerner A, Soudry M. Armed Conflict Injuries to the Extremities: A Treatment Manual. Springer Science & Business Media; 2011.
- [Background] Lundborg G. Nerve Injury and Repair: Regeneration, Reconstruction, and Cortical Remodeling. Elsevier/Churchill Livingstone; 2005.
- [Background] Brushart TM. Nerve Repair. Oxford University Press; 2011.
- [Background] Mackinnon SE, Dellon AL. Surgery of the Peripheral Nerve. Thieme Medical Publishers; 1988.
- [Background] Birch R. Surgical Disorders of the Peripheral Nerves. Springer London; 2011.
- [Background] Wilbourn AJ. The electrodiagnostic examination with peripheral nerve injuries. Clin Plast Surg. 2003 Apr;30(2):139-54. doi: 10.1016/s0094-1298(02)00099-8. PMID 12737349
- [Background] Seddon HJ, Medawar PB, Smith H. Rate of regeneration of peripheral nerves in man. J Physiol. 1943 Sep 30;102(2):191-215. doi: 10.1113/jphysiol.1943.sp004027. No abstract available. PMID 16991601
- [Background] SEDDON HJ. Nerve grafting. Ann R Coll Surg Engl. 1963 May;32(5):269-80. No abstract available. PMID 13987582
- [Background] SUNDERLAND S, BRADLEY KC. Denervation atrophy of the distal stump of a severed nerve. J Comp Neurol. 1950 Dec;93(3):401-9. doi: 10.1002/cne.900930304. No abstract available. PMID 14803568
- [Background] SUNDERLAND S. A classification of peripheral nerve injuries producing loss of function. Brain. 1951 Dec;74(4):491-516. doi: 10.1093/brain/74.4.491. No abstract available. PMID 14895767
- [Background] Sir SS. Nerves And Nerve Injuries. Churchill Livingstone; 1978
- [Background] Grass G, Kabir K, Ohse J, Rangger C, Besch L, Mathiak G. Primary Exploration of Radial Nerve is Not Required for Radial Nerve Palsy while Treating Humerus Shaft Fractures with Unreamed Humerus Nails (UHN). Open Orthop J. 2011;5:319-23. doi: 10.2174/1874325001105010319. Epub 2011 Aug 26. PMID 21915231
- [Background] Korompilias AV, Lykissas MG, Kostas-Agnantis IP, Vekris MD, Soucacos PN, Beris AE. Approach to radial nerve palsy caused by humerus shaft fracture: is primary exploration necessary? Injury. 2013 Mar;44(3):323-6. doi: 10.1016/j.injury.2013.01.004. Epub 2013 Jan 23. PMID 23352153
- [Background] Niver GE, Ilyas AM. Management of radial nerve palsy following fractures of the humerus. Orthop Clin North Am. 2013 Jul;44(3):419-24, x. doi: 10.1016/j.ocl.2013.03.012. Epub 2013 Apr 24. PMID 23827843
- [Background] Li Y, Ning G, Wu Q, Wu Q, Li Y, Feng S. Review of literature of radial nerve injuries associated with humeral fractures-an integrated management strategy. PLoS One. 2013 Nov 8;8(11):e78576. doi: 10.1371/journal.pone.0078576. eCollection 2013. PMID 24250799
- [Background] Rocchi M, Tarallo L, Mugnai R, Adani R. Humerus shaft fracture complicated by radial nerve palsy: Is surgical exploration necessary? Musculoskelet Surg. 2016 Dec;100(Suppl 1):53-60. doi: 10.1007/s12306-016-0414-3. Epub 2016 Nov 30. PMID 27900704
- [Background] Han SH, Hong IT, Lee HJ, Lee SJ, Kim U, Kim DW. Primary exploration for radial nerve palsy associated with unstable closed humeral shaft fracture. Ulus Travma Acil Cerrahi Derg. 2017 Sep;23(5):405-409. doi: 10.5505/tjtes.2017.26517. PMID 29052827
- [Background] Chang G, Ilyas AM. Radial Nerve Palsy After Humeral Shaft Fractures: The Case for Early Exploration and a New Classification to Guide Treatment and Prognosis. Hand Clin. 2018 Feb;34(1):105-112. doi: 10.1016/j.hcl.2017.09.011. PMID 29169591
- [Background] METRC Nerve Study: https://metrc.org/researchstudies/54-infopages/crsd/610-nervestudydescription - (personal communication, with interim results review performed in 3/2018).
- [Background] Perry JD. Electrodiagnosis in musculo-skeletal disease. Best Pract Res Clin Rheumatol. 2005 Jun;19(3):453-66. doi: 10.1016/j.berh.2005.01.007. PMID 15939369
- [Background] Korte N, Schenk HC, Grothe C, Tipold A, Haastert-Talini K. Evaluation of periodic electrodiagnostic measurements to monitor motor recovery after different peripheral nerve lesions in the rat. Muscle Nerve. 2011 Jul;44(1):63-73. doi: 10.1002/mus.22023. PMID 21674522
- [Background] Capacio BR, Byers CE, Matthews RL, Chang FC. A method for determining 4-aminopyridine in plasma: pharmacokinetics in anaesthetized guinea pigs after intravenous administration. Biomed Chromatogr. 1996 May-Jun;10(3):111-6. doi: 10.1002/(SICI)1099-0801(199605)10:33.0.CO;2-E. PMID 8792860
- [Background] Netter FH. Atlas of Human Anatomy, Professional Edition E-Book: including NetterReference.com Access with Full Downloadable Image Bank. Elsevier Health Sciences; 2014.
- [Background] Elfar JC, Yaseen Z, Stern PJ, Kiefhaber TR. Individual finger sensibility in carpal tunnel syndrome. J Hand Surg Am. 2010 Nov;35(11):1807-12. doi: 10.1016/j.jhsa.2010.08.013. PMID 21050964
- [Background] Sahin F, Atalay NS, Akkaya N, Ercidogan O, Basakci B, Kuran B. The correlation of neurophysiological findings with clinical and functional status in patients following traumatic nerve injury. J Hand Surg Eur Vol. 2014 Feb;39(2):199-206. doi: 10.1177/1753193413479507. Epub 2013 Mar 1. PMID 23456925
- [Background] Sims SE, Engel L, Hammert WC, Elfar JC. Hand Sensibility, Strength, and Laxity of High-Level Musicians Compared to Nonmusicians. J Hand Surg Am. 2015 Oct;40(10):1996-2002.e5. doi: 10.1016/j.jhsa.2015.06.009. Epub 2015 Aug 5. PMID 26253604
- [Background] Chimenti PC, McIntyre AW, Childs SM, Hammert WC, Elfar JC. Prospective cohort study of symptom resolution outside of the ulnar nerve distribution following cubital tunnel release. Hand (N Y). 2015 Jun;10(2):177-83. doi: 10.1007/s11552-014-9688-9. PMID 26034427
- [Background] Chimenti PC, McIntyre AW, Childs SM, Hammert WC, Elfar JC. Combined Cubital and Carpal Tunnel Release Results in Symptom Resolution Outside of the Median or Ulnar Nerve Distributions. Open Orthop J. 2016 May 24;10:111-9. doi: 10.2174/1874325001610010111. eCollection 2016. PMID 27347239
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Cohen J. A coefficient for agreement for nominal scales. Educational and Psychological Measurement. 1960;20:37-46.
- [Background] Fleiss JL. Measuring nominal scale agreement among many raters. Psychological Bulletin. 1971;76:378-382.
- [Background] Kim J, Farahmand M, Dunn C, Davies Z, Frisbee E, Milla C, Wine JJ. Evaporimeter and Bubble-Imaging Measures of Sweat Gland Secretion Rates. PLoS One. 2016 Oct 21;11(10):e0165254. doi: 10.1371/journal.pone.0165254. eCollection 2016. PMID 27768743
- [Background] Kiistala R, Kiistala U, Parkkinen MU, Mustakallio KK. Local sweat stimulation with the skin prick technique. Acta Derm Venereol. 1984;64(5):384-8. PMID 6208715
- [Background] Park SJ, Tamura T. Distribution of evaporation rate on human body surface. Ann Physiol Anthropol. 1992 Nov;11(6):593-609. doi: 10.2114/ahs1983.11.593. PMID 1476561
- [Background] Buchmann SJ, Penzlin AI, Kubasch ML, Illigens BM, Siepmann T. Assessment of sudomotor function. Clin Auton Res. 2019 Feb;29(1):41-53. doi: 10.1007/s10286-018-0530-2. Epub 2018 May 8. PMID 29737432
- [Background] Cardenas DD, Ditunno J, Graziani V, Jackson AB, Lammertse D, Potter P, Sipski M, Cohen R, Blight AR. Phase 2 trial of sustained-release fampridine in chronic spinal cord injury. Spinal Cord. 2007 Feb;45(2):158-68. doi: 10.1038/sj.sc.3101947. Epub 2006 Jun 13. PMID 16773037